CLINICAL TRIAL: NCT06265324
Title: Immediate and Midterm Clinical Outcome of Drug Coated Balloon Angioplasty in Different Coronary Artery Lesions in Sohag Governorate
Brief Title: Drug-coated Balloon Treatment in Coronary Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Imran Saber Mohamed, Assistant lecturer, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-12-04MD
Record Dates: First submitted 2024-02-04; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Drug-coated Balloon
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control (Experimental)
  Interventions: Device: Angioplasty

INTERVENTIONS:
Device: Angioplasty — Drug-coated balloons angioplasty for treatment of de novo and in-stent restenosis lesions

SUMMARY:
This study is multicenter registry for drug-coated balloon treatment for de novo and in-stent restenosis lesions

DETAILED DESCRIPTION:
The treatment of coronary lesions triggers processes in vessel walls with different characteristics depending on the revascularization strategy, post-traumatic healing following plain balloon angioplasty triggers vessel recoil and neointimal overgrowth, bare metal or drug eluting stent implantation results in neointimal cell proliferation, scar tissue formation, and ultimately, the generation of neoatherosclerosis Drug-coated balloons(DCBs) were presented two decades ago as an alternative to plain-balloon inﬂation or subsequent stent implantation in order to overcome in-stent restenosis.Recently, there has been growing evidence that DCBs can also be used off-label to treat de novo lesions in small vessels Therefore, the aim of this study is to evaluate efﬁcacy and safety of drug-coated balloons angioplasty for treatment of de novo and in-stent restenosis lesions

ELIGIBILITY:
Inclusion Criteria:

Eligible patients are those with lesions in the coronary vessel tree who will be planned to be treated with drug coated balloon.

Exclusion Criteria:

1. Severe renal impairment ( Cr.Cl. < 45 ml/min ).
2. Sever heart failure or liver cell failure .
3. Patients with contraindications to coronary angiography or invasive procedures.
4. Known allergy or intolerance to the medications or devices commonly used during PCI procedures.
5. Severe comorbidities or conditions that may limit life expectancy or impact the ability to follow the study protocol.
6. Pregnant or lactating women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2024-06-10 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events at 6 months | 6 months
  Primary endpoint is major adverse cardiac events (MACE is a composite of cardiac death, non-fatal myocardial infarction, target-vessel revascularization and major bleeding [BARC type 3 to 5]) at 6 months.
  1. Cardiac death: Any death due to proximate cardiac cause (eg, myocardial infarction, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure-related deaths, including those related to concomitant treatment, will be classified as cardiac death.
  2. Target vessel Revascularization: TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel.

CONTACTS AND LOCATIONS:
Overall Officials: Sharaf Eldin Shazly, PHD, Study Director — Sohag faculty of medicine; Mohammed Abdelwahab, PHD, Study Chair — Sohag faculty of medicine; Imran Saber, MA, Principal Investigator — Sohag faculty of medicine
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No